CLINICAL TRIAL: NCT05686564
Title: Early Access Program for ALXN1840 in Patients With Wilson Disease
Status: No longer available | Type: Expanded Access
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D9430R00001
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Wilson Disease
Keywords: Wilson Disease; ALXN1840
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: ALXN1840 — bis-choline tetrathiomolybdate
  Other Names: INN: tiomolibdic acid; USAN/JAN: tiomolibdate choline (WTX101)

SUMMARY:
This is an open-label, single-arm, multi-center EAP, designed to provide early access to ALXN1840 for eligible patients with WD.

DETAILED DESCRIPTION:
To provide access to ALXN1840 treatment, an investigational medicinal product (IMP) that has not yet been granted marketing authorization, to participants who complete Studies ALXN1840-WD-205, WTX101-301, or ALXN1840-WD-302, or other studies with ALXN1840 who, in the opinion of the Treating Physician, may benefit from continued treatment with ALXN1840, and who meet the eligibility criteria described in this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 3 years of age or older at the time of providing informed consent/assent and expressed desire to continue treatment with ALXN1840.
2. Confirmed diagnosis of WD.
3. Has completed one of the following ALXN1840 clinical studies:

   1. ALXN1840-WD-205
   2. WTX101-301
   3. ALXN1840-WD-302
   4. Other ALXN1840 studies
4. In the Treating Physician's medical opinion, the potential benefits of treatment with ALXN1840 outweigh the potential risks for the participant.
5. Participant or legal representative provided informed consent/assent to be treated with ALXN1840 through this EAP.
6. Female participants of childbearing potential and male participants must follow protocol-specified-contraception guidance.

Exclusion Criteria:

1. Eligible for and able to participate in an Alexion-sponsored study of ALXN1840.
2. Unwilling or unable to comply with the Treating Physician's treatment plan related to this EAP for any reason.
3. Has decompensated hepatic cirrhosis.
4. Model for End-Stage Liver Disease (MELD) score > 13.
5. Modified Nazer Score > 7.
6. End-stage renal disease on dialysis (chronic kidney disease stage 5 [CKD 5]) or creatinine clearance < 30 mL/min.
7. Known hypersensitivity to ALXN1840, ALXN1840 excipients, or any of the ingredients contained in ALXN1840.
8. Women who are nursing or pregnant (or women who are planning to become pregnant during treatment with ALXN1840).

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult